CLINICAL TRIAL: NCT04648163
Title: Suction Drain Volume Following Axillary Lymph Node Dissection for Malignant Melanoma - When to Remove Drains? A Retrospective Cohort Study.
Brief Title: Suction Drain in Axillary Lymph Node Dissection for Malignant Melanoma
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 29-607
Record Dates: First submitted 2020-11-04; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative complications like seroma formation and wound site infection readily occur following completion axillary lymph node dissection (ALND) for malignant melanoma. We analyzed the impact of time-to-drain removal and drainage volume on seroma formation after ALND.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed malignant melanoma
* underwent axillary lymph node dissection (level I-III)
* daily drainage volume records over a two-week period available

Exclusion Criteria:

* daily drainage volume records over a two-week period not available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Included patients had a histologically confirmed malignant melanoma (MM), underwent axillary lymph node dissection (level I-III) and had daily drainage volume records over a two-week period. Prior data collection we obtained ethical approval (institutional review board #25-438 ex 12/13). Data collection and analysis were performed in accordance with the rules set by the Declaration of Helsinki.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
daily drainage volume during hospitalization | through study completion, an average of 1 year
  The daily drainage amount durin hospital stay
total drainage volume during hospitalization | through study completion, an average of 1 year
  The total drainage amount during hospital stay
time-to-drain removal | through study completion, an average of 1 year
  The timepoint when the drain was removed
evacuation of seroma after drain removal | through study completion, an average of 1 year
  If evacuation of seroma after drain removal was needed

SECONDARY OUTCOMES:
demographic data - age | through study completion, an average of 1 year
  age
demographic data - sex | through study completion, an average of 1 year
  sex
demographic data - BMI | through study completion, an average of 1 year
  body mass index (BMI)
demographic data - smoking | through study completion, an average of 1 year
  smoking
demographic data - Diabetes mellitus | through study completion, an average of 1 year
  diabetes mellitus
demographic data - allergies | through study completion, an average of 1 year
  allergies
intraoperative parameters | through study completion, an average of 1 year
  surgical procedure time
intraoperative parameters - site | through study completion, an average of 1 year
  site
Amount of histologically analyzed lymph nodes | through study completion, an average of 1 year
  The amount lymph nodes found at histological analysis
Surgical complications | through study completion, an average of 1 year
  graded by the Clavien-Dindo-classification ( 1:normal postoperative cause without need of pharmacological treatment ; 2: pharmacological treatment ; 3: surgical, endoscooic or radiological treatment; 4: live-threating complications; 5: Death

CONTACTS AND LOCATIONS:
Overall Officials: David B Lumenta, MD, Prof, Study Chair — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria